CLINICAL TRIAL: NCT01680523
Title: A Randomized Controlled Trial Comparing Radical Hysterectomy Plus Tailored Adjuvant Therapy Versus Primary Chemoradiation Therapy in Bulky Early-stage Cervical Cancer (KGOG 1029)
Brief Title: Radical Hysterectomy Followed by Tailored Adjuvant Therapy Versus Primary Chemoradiation Therapy in Bulky Early-stage Cervical Cancer (KGOG 1029)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Hyun Nam, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KGOG 1029
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; bulky early-stage; locally advanced; radical hysterectomy; concurrent chemoradiation therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RH group (Experimental): Radical hysterectomy followed by tailored adjuvant therapy
  Interventions: Procedure: Radical hysterectomy; Radiation: Tailored adjuvant therapy
- CCRT group (Active Comparator): Primary concurrent chemoradiation therapy
  Interventions: Radiation: Primary chemoradiation therapy

INTERVENTIONS:
Procedure: Radical hysterectomy — Piver-Rutledge type III hysterectomy New classification type C2 hysterectomy Open, vaginal, laparoscopic assisted, laparoscopic, robotic radical hysterectomy are all allowed
  Arms: RH group
Radiation: Tailored adjuvant therapy — After radical hysterectomy, intermediate risk group according to GOG protocol 92 criteria will receive adjuvant radiation therapy. High risk group will receive adjuvant chemoradiation therapy with weekly cisplatin (40mg/m2, IV for 6 cycles). Extended filed radiation therapy is allowed in case of common iliac lymph node or para-aortic lymph node metastasis. Intracavitary brachytherapy and nodal or parametrial boost is not allowed.
  Other Names: Adjuvant radiation therapy; Adjuvant chemoradiation therapy
  Arms: RH group
Radiation: Primary chemoradiation therapy — Patient will receive primary radiation therapy including external pelvic irradiation, intracavitary brachytherapy, and parametrial or nodal boost. Extended filed radiation therapy is allowed in case of common iliac lymph node enlargement. Patients will receive concurrent weekly cisplatin (cisplatin 40mg/m2 for 6 cycles) during external radiation therapy.
  Arms: CCRT group

SUMMARY:
To compare 5-year overall survival between patients who undergo radical hysterectomy followed by tailored adjuvant therapy and patients who receive primary chemoradiation therapy in FIGO stage IB2 and IIA2 cervical cancer

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically confirmed cervical cancer
* FIGO stage IB2 and IIA2 disease
* One of following histologic types

  1. Squamous cell carcinoma
  2. Adenocarcinoma
  3. Adenosquamous carcinoma
* Gynecologic Oncology Group performance status: 0-2
* Adequate organ function

  1. Bone marrow: WBC > 3000/mm3, ANC ≥ 1,000/mm3, Platelet ≥ 100*103/mm3, Hemoglobin ≥ 10g/dL
  2. Kidney: Creatine < 1.25 * upper normal limit
  3. Liver: AST, ANT < 3 * upper normal limit, Total bilirubin < 1.5 mg/mm3
* Patient who have Singed an approved informed consent

Exclusion Criteria:

* Patients with cervical cancer who have received any previous radiation or chemotherapy
* Neuroendocrine carcinoma of uterine cervix
* Occult cervical cancer which was found after simple hysterectomy
* Para-aortic nodal involvement (> 10 mm short axis diameter on pretreatment imaging study)
* History of other invasive malignancies, with the exception of non-melanoma skin cancer, in situ melanoma and thyroid cancer, who had (or have) no evidence of the other cancer present within the last 5 years
* Serious illness or medical condition that precludes the safe administration of the trial treatment including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Prior diagnosis of Crohn's disease or ulcerative colitis
* Neurologic or psychiatric disease
* Patients who are pregnant or lactating

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Estimated)
Dates: Start 2012-09; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 year after treatment

SECONDARY OUTCOMES:
5-year progression-free survival | 5 years after treatment
Pattern of disease recurrence | within 5 years afer treatment
Treatment-related toxicity | within 5 years after treatment
  Treatment related toxicity will be evaluated using CTCAE v3.0.
Quality of life | within 1 year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hyun Nam, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea